CLINICAL TRIAL: NCT05156905
Title: A Phase 1b Trial Investigating Docetaxel Combined with Cirmtuzumab in Patients with Metastatic Castration Resistant Prostate Cancer
Brief Title: Study of Docetaxel Combined with Cirmtuzumab in Metastatic Castration Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Oncternal closing clinical trial operations.
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Rana Mckay, Associate Professor of Medicine and Urology, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-1514
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Prostate cancer; Docetaxel; Wnt pathway; Cirmtuzumab; ROR1
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cirmtuzumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cirmtuzumab + Docetaxel (Experimental): There is only one treatment arm on this study. The combination of cirmtuzumab + docetaxel will be administered on one treatment arm. Treatment will cirmtuzumab will be administered initially as a loading dose alone on days 1, 15, and 29 of cycle 1. Following the loading, cirmtuzumab will be given on Day 1 of every 21-day cycle starting on Cycle 2 to up to Cycle 7 corresponding with concurrent docetaxel administration. Following discontinuation or completion of docetaxel, treatment with cirmtuzumab will be continued Day 1 of every 28 cycle until disease progression, toxicity or study withdrawal. Docetaxel will be administered on day 1 of every 21-day cycle starting Cycle 2 for up to 6 cycles.
  Interventions: Drug: Cirmtuzumab

INTERVENTIONS:
Drug: Cirmtuzumab — Cirmtuzumab will be given in combination with docetaxel.
  Other Names: Docetaxel

SUMMARY:
The purpose of this study is to examine the safety and efficacy of cirmtuzumab in combination with standard of care docetaxel in patients with metastatic castration resistant prostate cancer. Docetaxel is a taxane chemotherapy which has been shown to prolong survival in men with castration resistant prostate cancer. Cirmtuzumab is a monoclonal antibody that targets the receptor called ROR1 of the non-canonical Wnt pathway and is suspected to contribute to prostate cancer growth and progression.

DETAILED DESCRIPTION:
This study seeks to targeting the non-canonical Wnt pathway with an antibody against ROR1. ROR1 is an attractive target given its low expression in non-malignant tissues and its role in proliferation and survival in prostate cancer. From preclinical data in a variety of tumor types, blockade of ROR1 inhibits cell growth and cirmtuzumab has shown efficacy in clinical trials with CLL. Preclinical data suggests that ROR1 is upregulated in chemotherapy resistant cells and treatment with cirmtuzumab and a taxane achieved higher cytotoxic response than both agents alone, supporting the use of the combination of cirmtuzumab and a taxane. Based on the biological rationale behind cirmtuzumab and preclinical activity with docetaxel, this is an open label, phase 2 clinical trial to evaluate the safety and efficacy of cirmtuzumab in combination with docetaxel for the treatment of metastatic, castrate resistant prostate adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically or cytologically confirmed adenocarcinoma of the prostate. Patients with neuroendocrine component are eligible.
2. Participants must have castrate levels of serum testosterone < 50 ng/dL.
3. Participants without orchiectomy must be maintained on luteinizing hormone releasing hormone (LHRH) agonist/antagonist.
4. Participants must have received prior abiraterone and/or next generation androgen receptor antagonist (enzalutamide, apalutamide, or darolutamide) for hormone sensitive disease or CRPC. Prior docetaxel for hormone sensitive disease is permitted.
5. Participants must have progressive disease. Patients with non-measurable disease are eligible.
6. Eastern Cooperative Oncology Group performance status ≤1 (Karnofsky ≥80%).
7. Patients must have normal organ and marrow function.

Exclusion Criteria:

1. No pure small cell carcinoma.
2. Prior treatment with cirmtuzumab.
3. No prior treatment with docetaxel for CRPC.
4. Treatment with abiraterone, apalutamide, or darolutamide within 2 weeks of treatment initiation. Treatment with cytotoxic chemotherapy within 3 weeks of treatment initiation. Treatment enzalutamide or other investigational prostate cancer directed therapy within 4 weeks of treatment initiation.
5. Palliative radiation therapy to the bone or other sites within 2 weeks of treatment initiation.
6. Imminent or established spinal cord compression based on clinical and/or imaging findings.
7. Known active central nervous system metastases and/or carcinomatous meningitis.
8. Uncontrolled intercurrent illness or clinically significant medical condition.
9. Treatment with antimicrobial agent within 4 weeks of treatment initiation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Recommended phase 2 dose of docetaxel combined with cirmtuzumab | Patients will be followed from study entry to death or date last known alive, assessed up to 36 months
  Defined by CTCAE version 5 grading

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events | Patients will be followed from study entry to death or date last known alive, assessed up to 36 months
  Defined by CTCAE version 5 grading
Total alkaline phosphatase response | Patients will be followed from study entry to death or date last known alive, assessed up to 36 months
  Defined as a reduction of ≥30% from the baseline value, confirmed ≥4 weeks later.
Time to PSA progression | Patients will be followed from study entry to death or date last known alive, assessed up to 36 months
  Defined by PCWG-3 criteria
Time to increase in the total alkaline phosphatase level | Patients will be followed from study entry to death or date last known alive, assessed up to 36 months
  Defined as an increase of ≥25% from baseline at ≥12 weeks, in patients with no decrease from baseline, or as an increase of ≥25% above the nadir, confirmed ≥3 weeks later, in patients with an initial decrease from baseline.
Radiographic progression free survival | Patients will be followed from study entry to death or date last known alive, assessed up to 36 months
  Defined by PCWG-3 criteria for bone metastases and RECIST version 1.1 for soft tissue
Time to first subsequent anti-cancer therapy | Patients will be followed from study entry to death or date last known alive, assessed up to 36 months
  Time from study discontinuation to initiation of subsequent systemic anti-cancer therapy or death
Time to first symptomatic skeletal event | Patients will be followed from study entry to death or date last known alive, assessed up to 36 months
  Time to first symptomatic pathologic fracture, radiation to the bone given symptomatic bone metastasis, surgery to the bone given symptomatic bone metastasis, or symptomatic spinal cord compression
Overall survival | Patients will be followed from study entry to death or date last known alive, assessed up to 36 months
  Time from enrollment to death or last follow up
Composite clinical benefit | Patients will be followed from study entry to death or date last known alive, assessed up to 36 months
  Composite endpoint of clinical benefit defined as any one of the following: PSA response by PCWG3 criteria, objective response rate by RECIST version 1.1, and stable disease > 6 months by RECIST version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Rana McKay, Study Chair — UCSD
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No